CLINICAL TRIAL: NCT01508130
Title: Non-Interventional, Prospective Cohort Study of the Effectiveness, Safety and Utilization of Two Approved Pegylated Interferon-Based Direct Acting Antiviral Triple Therapies in the Management of Genotype 1 Chronic Hepatitis C in Routine Clinical Practice in the USA
Brief Title: An Observational Study of Peginterferon (e.g. Pegasys)-Based Direct Acting Antiviral Triple Therapy in Patients With Chronic Hepatitis C Genotype 1
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27900
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will evaluate the efficacy and safety of two approved pegylated interferon-based direct acting antiviral triple therapies in patients with chronic hepatitis C genotype 1. Patients receiving pegylated interferon (e.g. Pegasys) and ribavirin plus either telaprevir or boceprivir in accordance with local standard of care and US labeling will be followed for the duration of their treatment and for up to 24 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic hepatitis C, genotype 1
* Receiving pegylated interferon-based direct acting antiviral therapy (pegylated interferon and ribavirin plus either telaprevir or boceprivir) in accordance with local standard of care and US labeling

Exclusion Criteria:

* Contraindications per US labels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C genotype 1 receiving pegylated interferon-based direct acting antiviral triple therapies in the US
Sampling Method: Probability Sample
Enrollment: 672 (Actual)
Dates: Start 2012-01-31 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (66):
- United States (65):
  - Cooper Green Hospital, Birmingham, Alabama
  - Univ. of Alabama at Birmingham; The Kirklin Clinic, Birmingham, Alabama
  - Liver Wellness Center, Little Rock, Arkansas
  - Loma Linda University Medical Center and Liver Center, Loma Linda, California
  - HMRI Liver Center, Pasadena, California
  - Kaiser Permanente San Diego; Hepatology Research, San Diego, California
  - VA San Diego Healthcare System, San Diego, California
  - South Bay Gastroenterology Medical Group, Torrance, California
  - University of Colorado Denver, Aurora, Colorado
  - Litchfield County Gastroenterology Associates, Torrington, Connecticut
  - Consultive Medicine, Daytona Beach, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - Center for Advanced Gastroenterology, Maitland, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Orlando Infectious Disease Center, Pa, Orlando, Florida
  - Tampa General Hospital; Tampa General Medical Group, Tampa, Florida
  - Atlanta Center for Gastroenterology, PC, Decatur, Georgia
  - Dekalb Gastroenterology Associates, Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - University of Chicago, Chicago, Illinois
  - Indianapolis Gastroenterology, Indianapolis, Indiana
  - Tristate Gastroenerology Associates, Crestview Hills, Kentucky
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - New Orleans Research Institute., Metairie, Louisiana
  - Tulane Uni Health Sciences Center, New Orleans, Louisiana
  - Mercy Medical Center; Institute For Digestive Health And Liver Disease, Baltimore, Maryland
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Baystate Infectious Diseases Clinical Research, Springfield, Massachusetts
  - Partners in Internal Medicine, Worcester, Massachusetts
  - Harper University Hospital/Wayne State, Detroit, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Midwest Biomedical Research Foundation, Kansas City, Missouri
  - Saint Louis University Gastroenterology & Hepatology; Clinical Research Unit, St Louis, Missouri
  - Dartmouth Hitchcock Med Center, Lebanon, New Hampshire
  - Lourdes Medical Associates; Southern New Jersey Center for LIver Disease, Haddon Heights, New Jersey
  - Atlantic Research Affiliates, Morristown, New Jersey
  - AGA Clinical Research Associates, LLC, Twp, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Mountainview Medical Practice, Catskill, New York
  - New Discovery, LLC, Flushing, New York
  - North Shore University Hospital, Manhasset, New York
  - Concorde Medical Group, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - Duke Univ Medical Center, Durham, North Carolina
  - Boice-Willis Clinic, Rocky Mount, North Carolina
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - DuBois Regional Medical Center, DuBois, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center; Division of Hepatology, Philadelphia, Pennsylvania
  - Methodist Heathcare University Hospital, Memphis, Tennessee
  - Imtiaz Alam MD, P.A. - Private Practice, Austin, Texas
  - Methodist Transplant Physicians, Dallas, Texas
  - Univ of Texas Medical Branch, Galveston, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Liver Associates of Texas, Houston, Texas
  - Digestive And Liver Disease Consultants, PA, Houston, Texas
  - University of Vermont, Burlington, Vermont
  - University of Virginia Health System: Gastroenterology at UVA, Charlottesville, Virginia
  - Metropolitan Research, Fairfax, Virginia
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 672 participants were enrolled at 64 study sites in the U.S between 20 January 2012 and 8 February 2013.
Pre-assignment Details: Out of 672 participants, one was not eligible to receive triple therapy (pegylated interferon alfa [PegIFN], ribavirin [RBV], and telaprevir or boceprevir) and 17 who received only dual therapy (PegIFN + RBV) were excluded from all analyses. A total of 635 participants were included in modified all treated (mTRT) population.
Groups:
- PegIFN + RBV + TEL: As per the standard of care and U.S. labeling, participants received PegIFN + RBV + telaprevir (TEL) for 12 weeks; followed by additional 12 or 36 weeks of PegIFN + RBV (dual therapy) depending on viral response and prior response status.
- PegIFN + RBV + BOC: As per the standard of care and U.S. labeling, participants received first 4 weeks of PegIFN + RBV (dual therapy), followed by additional 28 or 36 weeks of PegIFN + RBV + boceprevir (BOC) therapy, and/or then completed dual therapy through Week 48 depending on viral response and prior response status.
Period: Overall Study
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Started | 493 | 142
mTRT | 493 | 142
Completed | 266 | 73
Not Completed | 227 | 69
Not completed — Adverse Event | 81 | 28
Not completed — Death | 3 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 25 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Subject's substantial non-compliance | 25 | 9
Not completed — Insufficient therapeutic response | 74 | 23
Not completed — Administrative | 14 | 3

BASELINE CHARACTERISTICS:
Groups:
- PegIFN + RBV + TEL: As per the standard of care and U.S. labeling, participants received pegylated interferon alfa (PegIFN) + ribavirin (RBV) + telaprevir (TEL) for 12 weeks; followed by additional 12 or 36 weeks of PegIFN + RBV (dual therapy) depending on viral response and prior response status.
- Total: Total of all reporting groups
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC | Total
Number analyzed (Participants) | 493 | 142 | 635
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (10.3) | 51.6 (10.0) | 51.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 56 | 265
  Male | 284 | 86 | 370

OUTCOME MEASURES:

1. Primary Outcome: Time to Premature Treatment Discontinuation Due to Any Reason
Description: Time to premature treatment discontinuation for any reason (weeks) was calculated as follows: date of treatment discontinuation for any reason - first treatment administration date + 1/7. The estimated survivorship curves were obtained from Kaplan-Meier maximum likelihood estimates for each treatment group. Participants who completed the study treatment (including those who shorten the treatment based on response-guided therapy) were censored on their last dosing date.
Time Frame: Up to the treatment discontinuation or the date of the last dosing for participants who were ongoing or completed the study treatment (including those who shorten the treatment based on response-guided therapy)
Population: modified all-treated (mTRT) population: It included all enrolled participants who had an hepatitis C Virus Ribo Nucleic Acid (HCV RNA) of 50 IU/mL or more just prior to start chronic hepatitis C (CHC) therapy, received 1 triple therapy (PegIFN, RBV, and TEL or BOC), and treatment documentation was sufficient for assignment to treatment groups.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 493 | 142
weeks | 40.0 [34.0 to NA] — An upper limit of CI was non-estimable due to insufficient number of participants with events. | 40.6 [32.3 to 48.1]
Statistical Analysis 1: Comparison: PegIFN + RBV + TEL vs PegIFN + RBV + BOC; Test type: Superiority or Other; p = 0.6451, Wald residual chi-square test; Cox Proportional Hazard = 1.08, 95% CI 2-sided [0.78 to 1.49] — Due to the non-interventional study design, the Cox model included a propensity score as a covariate (incorporated important demographics and baseline characteristics) to account for the potential imbalance between treatment groups
Statistical Analysis 2: Comparison: PegIFN + RBV + TEL vs PegIFN + RBV + BOC; Test type: Superiority or Other; p = 0.8826, Wald residual chi-square test; Cox Proportional Hazard = 1.02, 95% CI 2-sided [0.78 to 1.34] — Without Propensity Score as a Covariate

2. Primary Outcome: Number of Participants With Sustained Virologic Response (SVR) at 12 Weeks or Later After Completion of the Treatment Period
Description: SVR rate defined as the number of participants with undetectable HCV RNA (i.e., HCV RNA less than 50 IU/mL) at 12 weeks or later post-completion of the treatment period
Time Frame: 12 weeks or later post-completion of the treatment period
Population: mTRT population: It included all enrolled participants with HCV RNA of 50 IU/mL or more just prior to start CHC therapy, received 1 triple therapy, and treatment documentation was sufficient for assignment to treatment groups.
Measure: Number; unit: participants
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 493 | 142
participants | 160 | 39
Statistical Analysis 1: Comparison: PegIFN + RBV + TEL vs PegIFN + RBV + BOC; Test type: Superiority or Other; p = 0.7695, Multiple Logistic Regression; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.58 to 1.49] — A multiple logistic regression model including a propensity score as a covariate (incorporated important demographics and baseline characteristics) was used for the treatment comparison
Statistical Analysis 2: Comparison: PegIFN + RBV + TEL vs PegIFN + RBV + BOC; Test type: Superiority or Other; p = 0.2594, Multiple Logistic Regression; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.84 to 1.92] — Without Propensity Score as a Covariate

3. Secondary Outcome: Number of Participants With Virologic Response (VR)
Description: VR was defined as undetectable HCV RNA (i.e.,HCV RNA less than 50 IU/mL)
Time Frame: Weeks 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48; and 12 weeks post-completion of treatment period
Population: mTRT population: It included all enrolled participants with HCV RNA of 50 IU/mL or more just prior to start CHC therapy, received 1 triple therapy, and treatment documentation was sufficient for assignment to treatment groups. "n" denotes number of participants who were available at the indicated time points for each arm.
Measure: Number; unit: participants
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 493 | 142
participants
  Week 2, n= 479, 138 | 104 | 3
  Week 4, n= 446, 137 | 348 | 19
  Week 6, n= 397, 128 | 327 | 33
  Week 8, n= 383, 125 | 349 | 87
  Week 12, n= 359, 113 | 337 | 102
  Week 16, n= 266, 91 | 244 | 86
  Week 20, n= 224, 80 | 209 | 75
  Week 24, n= 190, 70 | 176 | 67
  Week 28, n= 115, 29 | 105 | 26
  Week 32, n= 84, 23 | 78 | 20
  Week 36, n= 60, 16 | 56 | 14
  Week 40, n= 35, 10 | 33 | 9
  Week 44, n= 24, 6 | 23 | 5
  Week 48, n= 13, 1 | 13 | 1
  12 weeks post-completion, n= 187, 53 | 160 | 39

4. Secondary Outcome: Number of Participants With VR by Categories of Very Rapid VR (VRVR), Rapid Virological Response (RVR), VR Week 8, Early Virological Response (cEVR), Partial Virological Response (pEVR), and None of the Above
Description: VRVR was defined as HCV RNA < 50 IU/mL at treatment Week 2; RVR as HCV RNA < 50 IU/mL by treatment Week 4, but no HCV RNA < 50 IU/mL at Week 2; Week 8 VR as HCV RNA < 50 IU/mL by study Week 8 but no HCV RNA < 50 IU/mL at Weeks 2 to 4; cEVR as HCV RNA < 50 IU/mL by treatment Week 12 but no HCV RNA < 50 IU/mL at Weeks 2 to 8; and pEVR as at least a 2 log10 decrease in HCV RNA by treatment Week 12 but no HCV RNA < 50 IU/mL at Weeks 2 to 12.
Time Frame: Weeks 2, 4, 8, and 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 493 | 142
participants
  VRVR, Week 2, n= 479, 138 | 104 | 3
  RVR, Week 4, n= 446, 137 | 252 | 16
  VR Week 8, n= 383, 125 | 28 | 56
  cEVR, Week 12, n= 359, 113 | 17 | 18
  pEVR, Weeks 2 to 12, n= 359, 113 | 4 | 4
  None of above, Weeks 2 to 12, n= 359, 113 | 7 | 7

5. Secondary Outcome: Number of Participants Who Achieved Extended VR, Virologic Breakthrough/Rebound, Virologic Relapse, and Who Were Non-responder
Description: The extended VR is defined as initial HCV RNA < 50 IU/mL during Weeks 2 to 24 and remaining HCV RNA < 50 IU/mL at all subsequent assessments; virologic breakthrough/rebound is defined as detectable HCV RNA during the treatment period in participants with prior non-detectable HCV RNA or increase of HCV RNA by >=1 log10 above nadir for direct-acting antiviral (DAA) tripe therapies (PegIFN + RBV + TEL or PegIFN + RBV + BOC); virologic relapse is defined as detectable HCV RNA during the treatment-free follow-up period in participants with HCV RNA < 50 IU/mL at EoT; non-responder is defined as participants who never achieved undetectable HCV-RNA during the 48 weeks of treatment.
Time Frame: Up to Week 48
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 493 | 142
participants
  Extended VR, n= 491, 142 | 159 | 39
  Virologic breakthrough/rebound, n= 491, 142 | 52 | 15
  Virologic relapse, n= 491, 142 | 174 | 52
  Non-responders, n= 479, 138 | 34 | 16

6. Secondary Outcome: Predictors of Sustained Virologic Response by Week
Description: SVR rate defined as the number of participants with undetectable HCV RNA (i.e., HCV RNA less than 50 IU/mL) at 12 weeks or later post-completion of the treatment period. The predictors defined as participants with virological response (HCV RNA < 50 IU/mL at any visit), or with virological response at Week 12 (HCV-RNA < 50 IU/mL or unquantifiable or HCV-RNA >=2 log10 drop from baseline). Positive predictive value is the probability that participants with a positive screening test truly have the disease. Negative predictive value is the probability that participants with a negative screening test truly don't have the disease.
Time Frame: Weeks 2, 4, 6, 8, and 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 493 | 142
participants
  Week 2, positive predictors, n=104, 3 | 43 | 1
  Week 4, positive predictors, n=350, 19 | 138 | 10
  Week 6, positive predictors, n=336, 33 | 142 | 17
  Week 8, positive predictors, n=355, 88 | 147 | 33
  Week 12, positive predictors, n=348, 102 | 146 | 36
  VR, Week 12, positive predictors, n=347, 106 | 146 | 37
  Week 2, negative predictors, n=375, 135 | 258 | 97
  Week 4, negative predictors, n=96, 118 | 74 | 89
  Week 6, negative predictors, n=61, 95 | 50 | 74
  Week 8, negative predictors, n=28, 37 | 24 | 32
  Week 12, negative predictors, n=11, 11 | 11 | 9
  VR, Week 12, negative predictors, n=12, 7 | 12 | 6

7. Secondary Outcome: Number of Participants With SVR by Subgroups (Demographic and Baseline Factors)
Description: Participants for VR to prior therapy (PegIFN + RBV) were categorized as: relapse (who completed the previous treatment with HCV RNA undetectable, but relapsed with detectable HCV RNA once treatment was discontinued), breakthrough (HCV RNA undetectable, followed by detectable HCV RNA during on-treatment period), null responder (completed at least 12 weeks of treatment with HCV RNA decrease < 2 log10 at Week 12), partial responder (HCV RNA decrease > 2 log10 by Week 12 of treatment and HCV RNA remained detectable), unknown response (completed previous treatment, but treatment response based on HCV RNA determinations was not available), and prior intolerant (treated previously, but discontinued due to adverse event or participant's choice prior to completion of therapy). Participants categorized into 3 genotypes (CC, CT and TT) based on single nucleotide polymorphism in the Interleukin 28B (IL28B) gene.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 493 | 142
participants
  Sex : Female, n = 209, 56 | 76 | 22
  Sex: Male, n = 284, 86 | 84 | 17
  Age: < 50 years, n = 144, 47 | 49 | 14
  Age: >= 50 years, n = 349, 95 | 111 | 25
  Race: White, n = 336, 102 | 112 | 31
  Race: non-white, n = 157, 40 | 48 | 8
  Ethnicity: Hispanic or Latino, n = 42, 11 | 21 | 2
  Ethnicity: Not Hispanic or Latino, n = 450, 128 | 139 | 36
  Ethnicity: Unknown, n = 1, 3 | 0 | 1
  HCV Genotype: 1a, n = 350, 94 | 109 | 28
  HCV Genotype: 1b, n = 96, 30 | 43 | 7
  HCV Genotype: Other(2,3,4) , n = 45, 17 | 7 | 4
  HCV Genotype: missing, n = 2, 1 | 1 | 0
  IL28B Genotype: CC, n = 37, 12 | 17 | 6
  IL28B Genotype: CT, n = 85, 31 | 28 | 8
  IL28B Genotype: TT, n = 24, 6 | 5 | 1
  IL28B Genotype: not available, n = 347, 93 | 110 | 24
  VR to Prior Therapy: relapser, n = 64, 21 | 26 | 7
  VR to Prior Therapy: breakthrough, n = 3, 2 | 2 | 1
  VR to Prior Therapy: null responder, n = 62, 10 | 11 | 1
  VR to Prior Therapy: partial responder, n = 29, 7 | 8 | 1
  VR to Prior Therapy: unknown response, n = 21, 1 | 11 | 0
  VR to Prior Therapy: prior intolerant, n = 22, 14 | 5 | 1
  VR to Prior Therapy: missing, n = 291, 87 | 97 | 28

8. Secondary Outcome: Duration of Viral Undetectability During Treatment for Participants With HCV RNA Undetectable During Treatment by Trial Treatment
Description: The undetectable HCV RNA means HCV RNA values less than 50 IU/mL. This outcome measure was calculated as the duration of participant's first date of undetectable HCV RNA and the date of the participant's last dose.
Time Frame: Up to Week 48
Population: as for outcome 2
Measure: Median (Full Range); unit: weeks
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 159 | 39
weeks | 22.1 [0 to 52] | 23.0 [5 to 44]

9. Secondary Outcome: Time to Premature Treatment Discontinuation Due to Lack of Efficacy
Description: The participants discontinued the study treatment due to lack of efficacy of study treatment. Time to premature treatment discontinuation due to lack of efficacy (weeks) = (date of treatment discontinuation due to lack of efficacy - first treatment administration date + 1)/7. Participants who were ongoing or completed the study treatment (including those who shortened the treatment based on response-guided therapy) were censored at the date of their last dosing.
Time Frame: Up to Week 48
Population: as for outcome 2
Measure: Median (Full Range); unit: Weeks
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 493 | 142
Weeks | NA [0.1 to 64.3] — Median was non-estimable due to insufficient number of participants with premature treatment discontinuation. | NA [3.9 to 50.7] — Median was non-estimable due to insufficient number of participants with premature treatment discontinuation.
Statistical Analysis 1: Comparison: PegIFN + RBV + TEL vs PegIFN + RBV + BOC; Test type: Superiority or Other; p = 0.9156, Wald residual chi-square test; Cox Proportional Hazard = 1.03, 95% CI 2-sided [0.64 to 1.64] — 95% CI for median was computed using the method of Brookmeyer and Crowley

10. Secondary Outcome: Time to Premature Treatment Discontinuation Due to Intolerance
Description: The participants discontinued the study treatment due to intolerance of the study treatment. Time to premature treatment discontinuation due to intolerance (weeks) = (date of treatment discontinuation due to lack of intolerance - first treatment administration date + 1)/7. Participants who were ongoing or completed the study treatment (including those who shortened the treatment based on response-guided therapy) were censored at the date of their last dosing.
Time Frame: Up to Week 48
Population: as for outcome 2
Measure: Median (Full Range); unit: Weeks
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 493 | 142
Weeks | NA [0.1 to 64.3] — Median was non-estimable due to insufficient number of participants with premature treatment discontinuation. | NA [3.9 to 50.7] — Median was non-estimable due to insufficient number of participants with premature treatment discontinuation.
Statistical Analysis 1: Comparison: PegIFN + RBV + TEL vs PegIFN + RBV + BOC; Test type: Superiority or Other; p = 0.5649, Wald residual chi-square test; Cox Proportional Hazard = 0.88, 95% CI 2-sided [0.57 to 1.36] — 95% CI for median was computed using the method of Brookmeyer and Crowley

11. Secondary Outcome: Treatment Duration, as Measure of Extent of Exposure to Study Medication
Description: Extent of exposure is defined as the duration of the treatment administered during the study. The mean duration of exposure to PegIFN alfa-2a, PegIFN alfa-2b, ribavirin, telaprevir, and boceprevir is calculated as the number of weeks between the start and end of treatment.
Time Frame: From the date of the first dose of the study drug up to withdrawal/study completion (up to Study Week 48)
Population: Safety population: It included all enrolled participants who received at least one dose of study treatment (triple therapy) and had at least one post-baseline safety assessment. "n" denotes number of participants who were available at the indicated time points for each arm.
Measure: Mean (Standard Error); unit: Weeks
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 490 | 142
Weeks
  PegIFN alfa-2a, n = 465, 127 | 26.0 (0.71) | 26.8 (1.16)
  PegIFN alfa-2b, n = 28, 15 | 23.2 (2.58) | 34.0 (3.12)
  Ribavirin, n = 490, 142 | 26.1 (0.69) | 27.6 (1.11)
  Telaprevir, n = 490, NA | 13.4 (0.39) | NA (NA) — Not applicable for this group.
  Boceprevir, n = NA, 142 | NA (NA) — Not applicable for this group. | 22.1 (1.07)

12. Secondary Outcome: Mean Cumulative Dose, as Measure of Extent of Exposure to Study Medication
Description: Extent of exposure is defined as the duration of the treatment administered during the study. The mean cumulative doses of PegIFN alfa-2a, PegIFN alfa-2b, ribavirin, telaprevir, and boceprevir were presented.
Time Frame: From the date of the first dose of the study drug up to withdrawal/study completion (up to Study Week 48)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 490 | 142
Micrograms
  PegIFN alfa-2a, n = 465, 127 | 4504.5 (2679.7) | 4478.1 (2275.6)
  PegIFN alfa-2b, n = 28, 15 | 3234.5 (2008.5) | 4239.1 (1723.5)
  Ribavirin, n = 490, 142 | 24991.1 (16058.1) | 26215.9 (14292.7)
  Telaprevir, n = 490, NA | 29734.2 (18776.5) | NA (NA) — Not applicable for this group.
  Boceprevir, n = NA, 142 | NA (NA) — Not applicable for this group. | 52979.7 (30728.6)

13. Secondary Outcome: Percentage of Dose Reduction, as Measure of Extent of Exposure to Study Medication
Description: Extent of exposure is defined as the duration of the treatment administered during the study. Degree of dose reduction was calculated as actual exposure/target exposure × 100%. Target exposure was defined as the actual received treatment duration multiplied by the initial assigned dose. Actual exposure was defined as cumulative dose during the treatment period.
Time Frame: From the date of the first dose of the study drug up to withdrawal/study completion (up to Study Week 48)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage of dose reduction
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 490 | 142
Percentage of dose reduction
  PegIFN alfa-2a, n = 465, 127 | 102.5 (10.1) | 104.8 (15.5)
  PegIFN alfa-2b, n = 28, 15 | 101.2 (6.0) | 111.7 (23.6)
  Ribavirin, n = 490, 142 | 116.8 (26.6) | 118.2 (25.6)
  Telaprevir, n = 490, NA | 100.0 (0.00) | NA (NA) — Not applicable for this group.
  Boceprevir, n = NA, 142 | NA (NA) — Not applicable for this group. | 99.8 (1.9)

14. Secondary Outcome: Compliance of Study Treatment
Description: Compliance was assessed based on the number of participants who received the planned study treatment (PegIFN alfa-2a, PegIFN alfa-2b, ribavirin, telaprevir, and boceprevir) during the treatment period.
Time Frame: Weeks 4, 8, 12, and 24
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 490 | 142
participants
  PegIFN Week 4; n = 345, 114 | 342 | 113
  PegIFN Week 8; n = 319, 107 | 312 | 103
  PegIFN Week 12; n = 310, 106 | 304 | 101
  PegIFN Week 24; n = 265, 88 | 259 | 83
  Ribavirin Week 4; n = 337, 111 | 331 | 105
  Ribavirin Week 8; n = 293, 101 | 281 | 100
  Ribavirin Week 12; n = 288, 98 | 279 | 93
  Ribavirin Week 24; n = 187, 77 | 180 | 69
  Telaprevir Week 4; n = 340, NA | 329 | NA — Not applicable for this group.
  Telaprevir Week 8; n = 309, NA | 289 | NA — Not applicable for this group.
  Telaprevir Week 12; n = 273, NA | 255 | NA — Not applicable for this group.
  Telaprevir Week 24; n = 68, NA | 67 | NA — Not applicable for this group.
  Boceprevir Week 4; n = NA, 34 | NA — Not applicable for this group. | 33
  Boceprevir Week 8; n = NA, 103 | NA — Not applicable for this group. | 93
  Boceprevir Week 12; n = NA, 101 | NA — Not applicable for this group. | 89
  Boceprevir Week 24; n = NA, 82 | NA — Not applicable for this group. | 70

15. Secondary Outcome: Number of Participants Treated With PegIFN, RBV, and TEL as Per the U.S. Label
Description: As per the U.S. labeling, participants with treatment-naive, prior relapse (TN-PR) and prior partial or null responder (PP/NR) received PegIFN + RBV + TEL (triple therapy) for 12 weeks; followed additional 12 or 36 weeks of PegIFN + RBV (dual therapy) depending on viral response and prior response status.
Time Frame: Up to 48 weeks (included 12 weeks of triple therapy + additional 12/36 weeks of dual therapy)
Population: as for outcome 11
Measure: Number; unit: participants
Groups:
- PegIFN + RBV + TEL: As per the standard of care and U.S. labeling, participants received first 4 weeks of PegIFN + RBV (dual therapy), followed by additional 28 or 36 weeks of PegIFN + RBV + boceprevir (BOC) therapy, and/or then completed dual therapy through Week 48 depending on viral response and prior response status.
Arm/Group | PegIFN + RBV + TEL
Number analyzed (Participants) | 490
participants
  TN-PR, 12 weeks, n = 352 | 190
  TN-PR, additional 12 weeks, n = 352 | 75
  TN-PR, additional 36 weeks, n = 352 | 8
  PP/NR, 12 weeks, n = 90 | 58
  PP/NR, additional 36 weeks, n = 90 | 25

16. Secondary Outcome: Number of Participants Treated With PegIFN, RBV, and BOC as Per the U.S. Label
Description: As per the U.S. labeling, participants with cirrhosis (C); non-cirrhotic/treatment-naïve (NC/TN); and non-cirrhotic/previous partial responders or relapsers (NC/PPR or R) received first 4 weeks of dual therapy, followed by additional 28 or 36 weeks of PegIFN + RBV + BOC (triple therapy) and/or then completed dual therapy through Week 48 depending on viral response and prior response status.
Time Frame: Up to 48 weeks (included 4 weeks of dual therapy + additional 28/36 weeks of triple therapy and/or additional dual therapy up to Week 48)
Population: The safety population was defined as all enrolled participants who received at least one dose of study treatment (triple therapy) and had at least one post-baseline safety assessment. "n" denotes number of participants who were available at the indicated time points for each arm.
Measure: Number; unit: participants
Arm/Group | PegIFN + RBV + BOC
Number analyzed (Participants) | 142
participants
  NC/TN, 4 weeks, n = 60 | 59
  NC/TN, additional 28 weeks, n = 24 | 15
  NC/TN, additional 36 weeks, n = 7 | 1
  NC/TN, dual therapy through 48 week, n = 7 | 2
  NC/PPR or R, 4 weeks, n = 17 | 17
  NC/PPR, additional 36 weeks, n = 7 | 3
  NC/PPR, dual therapy through 48 week, n = 3 | 1
  C, completed 44 weeks, n = 34 | 1

17. Secondary Outcome: Number of Participants With Safety-related Dose Reductions
Description: The dose reduction was done because of safety-related reasons (AEs) including alanine aminotransferase disorder, anemia, neutropenia, thrombocytopenia, and rash.
Time Frame: Up to 48 weeks
Population: Safety population: It included all enrolled participants who received at least one dose of study treatment (triple therapy) and had at least one post-baseline safety assessment.
Measure: Number; unit: participants
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 490 | 142
participants | 190 | 70

18. Secondary Outcome: Number of Participants With Premature Treatment Discontinuation Due to Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product.
Time Frame: Up to 48 weeks
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 490 | 142
participants | 80 | 28

19. Secondary Outcome: Number of Participants With Any AEs and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: Up to 12 weeks post-treatment
Population: Safety population: It included all enrolled participants who received at least one dose of study treatment (triple therapy) and had at least one post-baseline safety assessment. All 671 participants received at least one dose of study drug; however, 632 of these participants were included in the safety population.
Measure: Number; unit: participants
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 490 | 142
participants
  Any AEs | 470 | 142
  Any SAEs | 76 | 16

20. Secondary Outcome: Change From Baseline in Work Loss And Productivity Outcomes (WPAI)
Description: WPAI-AS is a 6-question participant rated questionnaire to determine the amount of absenteeism, presenteeism, work productivity loss and daily activity impairment attributable to ankylosing spondylitis for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism or reduced on-the-job effectiveness), overall work impairment (work productivity loss or absenteeism plus presenteeism) and activity impairment (daily activity impairment). Each sub-scores was scaled as 0 (not affected/no impairment) to 10 (completely affected/impaired). Higher scores indicated greater impairment and less productivity.
Time Frame: Baseline (Day 1 ), Weeks 2, 4, 6, 8, 12, 16, 24, 36, 48, 12 weeks post-treatment
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Number analyzed (Participants) | 493 | 142
units on a scale
  Wk 2, Work Time Missed, n = 37, 7 | 14.6 (3.09) | 13.8 (6.98)
  Wk 2, Impairment While Working (n = 36, 8) | 9.3 (3.79) | 19.6 (8.18)
  Wk 2, Overall work impairment (n = 35, 7) | 11.8 (4.31) | 26.8 (9.91)
  Wk 2, Activity impairment (n = 93, 33) | 16.7 (2.75) | 16.0 (4.63)
  Wk 4, Work Time Missed (n = 58, 16) | 10.8 (3.68) | 13.2 (7.07)
  Wk 4, Impairment While Working (n = 55, 16) | 21.8 (3.89) | 20.1 (7.28)
  Wk 4, Overall work impairment (n = 55, 16) | 25.3 (4.25) | 22.6 (7.95)
  Wk 4, Activity impairment (n = 142, 49) | 23.0 (2.73) | 11.5 (4.67)
  Wk 6, Work Time Missed (n = 25, 4) | 10.8 (4.34) | 31.0 (11.14)
  Wk 6, Impairment While Working (n = 25, 4) | 25.5 (6.36) | 0.6 (16.40)
  Wk 6, Overall work impairment (n = 25, 4) | 32.9 (6.02) | 24.7 (15.46)
  Wk 6, Activity impairment (n = 75, 29) | 17.9 (3.76) | 21.9 (6.10)
  Wk 8, Work Time Missed (; n = 48, 10) | 24.1 (5.03) | 0.2 (11.50)
  Wk 8, Impairment While Working (n = 45, 11) | 29.1 (3.77) | 7.1 (7.88)
  Wk 8, Overall work impairment (n = 44, 10) | 37.1 (4.15) | 7.5 (9.13)
  Wk 8, Activity impairment (n = 109, 40) | 30.7 (3.20) | 21.2 (5.32)
  Wk 12, Work Time Missed (n = 50, 11) | 17.6 (4.72) | -3.7 (10.24)
  Wk 12, Impairment While Working (n = 46, 10) | 28.2 (4.39) | 9.5 (9.57)
  Wk 12, Overall work impairment (n = 46,11) | 34.1 (4.43) | 2.8 (9.25)
  Wk 12, Activity impairment (n = 119, 41) | 27.3 (2.99) | 20.8 (5.12)
  Wk 16, Work Time Missed (n = 31, 10) | 1.5 (5.56) | 7.4 (10.11)
  Wk 16, Impairment While Working (n = 32, 10) | 21.0 (5.94) | 19.9 (11.0)
  Wk 16, Overall work impairment (n = 31, 10) | 23.9 (6.43) | 16.1 (11.69)
  Wk 16, Activity impairment (n = 87, 36) | 22.7 (3.90) | 19.7 (6.11)
  Wk 24, Work Time Missed (n = 22, 7) | 2.9 (5.09) | 17.0 (9.32)
  Wk 24, Impairment While Working (n = 21, 7) | 18.1 (8.35) | 11.5 (15.01)
  Wk 24, Overall work impairment (n = 21, 7) | 16.0 (7.59) | 25.3 (13.64)
  Wk 24, Activity impairment (n = 75, 35) | 14.5 (3.97) | 13.0 (5.83)
  Wk 36, Work Time Missed (n = 10, 1) | 2.8 (6.74) | 9.5 (26.28)
  Wk 36, Impairment While Working (n = 9, 1) | 14.4 (12.91) | 40.0 (47.92)
  Wk 36, Overall work impairment (n = 10, 1) | 13.5 (14.16) | 34.1 (55.23)
  Wk 36, Activity impairment (n = 28, 8) | 16.2 (6.21) | 10.9 (12.04)
  Wk 48, Work Time Missed (n = 4, 1) | 3.6 (50.76) | 119.0 (181.99)
  Wk 48, Impairment While Working (n = 3, 1) | 71.8 (52.43) | -5.4 (145.43)
  Wk 48, Overall work impairment (n = 4, 1) | 71.8 (48.32) | -67.1 (173.24)
  Wk 48, Activity impairment (n = 8, 1) | 35.4 (14.41) | 37.1 (59.10)
  EOT visit, Work Time Missed (n = 49, 10) | 8.4 (3.20) | 5.0 (7.30)
  EOT visit, Impairment While Working (n = 47, 10) | 20.8 (4.10) | 15.5 (9.15)
  EOT visit, Overall work impairment (n = 48, 10) | 24.2 (4.45) | 16.2 (10.04)
  EOT visit, Activity impairment (n = 143, 44) | 18.7 (2.97) | 14.8 (5.43)
  12 Wks in FU, Work Time Missed (n = 19, 3) | 16.8 (8.11) | -32.6 (21.41)
  12 Wks in FU, Impairment While Working (n = 19, 3) | 1.5 (3.51) | 3.6 (9.50)
  12 Wks in FU, Overall work impairment (n = 18, 3) | 13.6 (9.17) | -24.5 (24.09)
  12 Wks in FU, Activity impairment (n = 67, 17) | 0.8 (3.86) | -11.5 (7.66)

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: SAEs and other AEs were collected in the safety population, which was defined as all enrolled participants who received at least one dose of study treatment (triple therapy) and had at least one post-baseline safety assessment
Arm/Group | PegIFN + RBV + TEL | PegIFN + RBV + BOC
Serious Adverse Events (participants affected / at risk) | 76/490 | 16/142
Other Adverse Events (participants affected / at risk) | 470/490 | 142/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PegIFN + RBV + TEL (N=490) | PegIFN + RBV + BOC (N=142)
Pneumonia (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Wound infection (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Fungal sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 11 | 3
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal (Gastrointestinal disorders) | 1 | 0
Hemorrhage Vomiting (Gastrointestinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 4 | 0
Hepatic encephalopathy (Nervous system disorders) | 2 | 1
Migraine (Nervous system disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Cyst (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 2
Completed suicide (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Anticoagulation drug level below therapeutic (Investigations) | 1 | 0
Urine output decreased (Investigations) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PegIFN + RBV + TEL (N=490) | PegIFN + RBV + BOC (N=142)
Influenza-like illness (Infections and infestations) | 32 | 21
Anemia (Blood and lymphatic system disorders) | 249 | 87
Nausea (Gastrointestinal disorders) | 173 | 58
Diarrhoea (Gastrointestinal disorders) | 102 | 28
Decreased appetite (Gastrointestinal disorders) | 67 | 21
Vomiting (Gastrointestinal disorders) | 59 | 18
Anorectal discomfort (Gastrointestinal disorders) | 72 | 2
Constipation (Gastrointestinal disorders) | 44 | 12
Abdominal pain (Gastrointestinal disorders) | 40 | 11
Anal pruritus (Gastrointestinal disorders) | 33 | 3
Dyspepsia (Gastrointestinal disorders) | 29 | 5
Headache (Nervous system disorders) | 93 | 36
Dizziness (Nervous system disorders) | 70 | 28
Dysgeusia (Nervous system disorders) | 23 | 35
Paraesthesia (Nervous system disorders) | 38 | 2
Disturbance in attention (Nervous system disorders) | 32 | 7
Hypoaesthesia (Nervous system disorders) | 34 | 4
Fatigue (General disorders) | 265 | 82
Pyrexia (General disorders) | 69 | 15
Chills (General disorders) | 59 | 14
Insomnia (Psychiatric disorders) | 125 | 29
Depression (Psychiatric disorders) | 83 | 28
Irritability (Psychiatric disorders) | 56 | 21
Anxiety (Psychiatric disorders) | 48 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 102 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 71 | 23
Asthenia (Respiratory, thoracic and mediastinal disorders) | 72 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 25 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 170 | 23
Rash (Skin and subcutaneous tissue disorders) | 99 | 17
Rash pruritic (Skin and subcutaneous tissue disorders) | 65 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 54 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 27 | 13
Neutropenia (Investigations) | 58 | 32
Thrombocytopenia (Investigations) | 60 | 18
Leukopenia (Investigations) | 23 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 71 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 | 10
Vision blurred (Eye disorders) | 39 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.